CLINICAL TRIAL: NCT02111772
Title: Evaluating the Asthmatic Response to an Experimental Infection With Rhinovirus in the Atopic Host
Brief Title: Evaluating the Asthmatic Response to an Experimental Infection With Rhinovirus in the Atopic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Peter Heymann, MD, Head Pediatric Allergy and Immunology, University of Virginia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 12673; R01AI020565 (NIH)
Record Dates: First submitted 2014-03-27; First posted 2014-04-11 (Estimated); Results first posted 2018-05-29 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Asthma
Keywords: mild asthma, rhinovirus, young adults
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Asthmatic subjects (Experimental): Subjects with Asthma whose cold and chest symptoms will be evaluated one week before and 4 weeks after an inoculation with rhinovirus.
  Interventions: Biological: Rhinovirus
- Without Asthma (Active Comparator): Subjects without asthma whose cold and chest symptoms will be evaluated one week before and 4 weeks after an inoculation with rhinovirus
  Interventions: Biological: Rhinovirus

INTERVENTIONS:
Biological: Rhinovirus

SUMMARY:
In patients with asthma, reactions to allergens in the environment (such as mold, pollen, weed, domestic pets, and dust allergens) play an important role in causing asthma symptoms. However, upper respiratory tract infections, typically those caused by the common cold virus, rhinovirus, can also cause asthma to get worse. In previous studies at the University of Virginia, it was found that mild asthmatics, who had high levels of the allergy antibody (called IgE) in their blood, developed more persistent cold and chest symptoms when they were given an infection with rhinovirus (the most frequent cause of the common cold). The cold symptoms produced by rhinovirus tend to peak during the first 4 -7 days of the cold. These symptoms, including nasal congestion, are similar to what you have experienced with previous colds.

This study is being done to learn how a common cold caused by a viral infection affects people with asthma. The goal is to learn how to improve the care of asthma symptoms caused by the common cold virus (called rhinovirus). Most adults experience one or two colds caused by rhinovirus every year. In addition, 75-80% of asthma exacerbations caused by viral infections are caused by this virus, primarily in children. Adults are less likely to experience significant changes in their asthma symptoms when they get colds, because they have developed protective immune responses from previous colds which help diminish symptoms.

DETAILED DESCRIPTION:
Using rhinovirus strain 16 (RV-16) for inoculation, this study is designed to examine mechanisms of the asthmatic response to RV in the atopic host. In keeping with this, the primary objective of this investigation will be to test the hypothesis that mild asthmatics enrolled in this study will experience significantly increased lower respiratory tract symptoms over the first 4 days after experimental inoculation with RV-16 than non-allergic, non-asthmatic controls (as shown in our previous studies). It is anticipated that the results will serve to guide the development of new treatments to prevent asthma attacks provoked by RV. This will be a 5 week longitudinal study of 18 young allergic adults with mild asthma and 18 non-asthmatic controls who will be evaluated for 1 week to establish baseline symptoms and lung function, followed by an inoculation with rhinovirus (strain-16) and subsequent clinical and laboratory (mechanistic) monitoring for an additional 4 weeks. To participate in this study, subjects must live within 90 minutes by car from the University of Virginia.

Note: This study has been reviewed and is being monitored for safety by the NIH/NIAID Safety Monitoring Committee and by teh University of Virginia IRB (#12673). The virus pool used for inoculation has been produced under GMP conditions and is approved for this research by the FDA.

ELIGIBILITY:
Inclusion Criteria • ALL SUBJECTS:

* Subjects must be able to understand and provide written informed consent
* Age 18 to < 40 years of age, any gender, any racial/ethnic origin.
* Participant must be willing to comply with study procedures and requirements. Participant must be considered eligible for participation based on results of screening procedures conducted by protocol number 20100686 at VCU and IRB# 12656 at UVA.

Subjects with asthma

Criteria for inclusion will include those:

* with physician-diagnosed, mild asthma who are only using bronchodilators (e.g. albuterol) for symptom control.
* Asthma Control Test (ACT) Questionnaire Score a > 19 at enrollment (See Appendix: Asthma Control Test).
* Short-acting beta-agonist use < daily in last 4 weeks
* FEV1 > 70%, or FEV1/FVC ratio > 75% for subjects with FVC values between 80 and 87% predicted whose FEV1 values fall below 70%. a positive methacholine challenge test (i.e. at least a 20% fall in FEV1) at a methacholine concentration of 16 mg/ml or less (15). The methacholine test will not be done if subjects have used albuterol within 4 hours of the test procedure.Evidence for atopy demonstrated during screening (under IRB protocol# 12656) as judged by positive prick skin tests to one or more aero-allergens.

Control subjects. Criteria for inclusion will include those who do not have a history of asthma or allergic disorders (e.g. allergic rhinitis, atopic dermatitis, or food allergies).

Exclusion Criteria ALL SUBJECTS:

* Inability or unwillingness of a participant or subject's legal representative to give written informed consent and HIPPA authorization
* Positive test for serum neutralizing antibody to RV-16. Subjects with a neutralizing antibody titer > 1:4 will be excluded.
* Chronic heart disease, lung diseases other than asthma, or other chronic illnesses, including primary and/or secondary immunodeficiency.
* An upper or lower respiratory tract infection within six weeks prior to enrollment
* Who have required nasal or sinus surgery, excluding surgery for a deviated septum within 12 months prior to enrollment.
* Who have a 5 pack/year history of smoking, or any smoking within the last 6 months.
* Female subjects who are or who plan to become pregnant during the study, or who are nursing a baby. Additionally, to be included in this study, a woman of child-bearing potential must have a negative urine pregnancy test at screening, during the run-in, and prior to viral inoculation and agree to use an effective method of birth control such as, but not limited to, birth control pills, contraceptive foam, diaphragm, IUD, abstinence, or condoms.
* Absolute neutrophil count (ANC) < 1800 cells/mm3 (or 1.8 K/uL) detected during screening within 6 weeks of enrollment.

Subjects with asthma

Criteria for exclusion will include those:

* Who have required inhaled steroids (used for asthma), nasal steroids (used for allergic rhinitis), cromolyn, nedocromil sodium, ipratropium bromide, or leukotriene modifiers during the month prior to enrollment, oral steroids within 6 weeks of enrollment, omalizumab (Xolair®) within 12 months prior to enrollment, or who are currently using beta adrenergic blocking agents.
* Who have been hospitalized or treated in the emergency room (unless the treatment involved the use of a bronchodilator only) for asthma within the last three years.
* To avoid RV-16 inoculations in subjects with more restrictive lung volumes, those whose FVC is < 80% predicted will be excluded. Subjects who are currently receiving allergen immunotherapy (IT), or who have received allergen IT within the last 3 years.
* Subjects who have had one or more night time awakenings caused by asthma symptoms and/or who have needed their SABA (albuterol) inhaler for asthma symptoms > 4 days during the week before enrollment, or during the week before the inoculation with RV-16.

Control subjects

• Who have a positive methacholine test, or positive prick skin tests at screening under IRB protocol # 12656.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2013-09-01; Primary Completion 2017-04-20 (Actual); Study Completion 2017-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heymann W Peter, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Asthmatic Subjects: Subjects with Asthma whose cold and chest symptoms will be evaluated one week before and 4 weeks after an inoculation with rhinovirus.
  Rhinovirus
- Without Asthma: Subjects without asthma whose cold and chest symptoms will be evaluated one week before and 4 weeks after an inoculation with rhinovirus
  Rhinovirus
Period: Overall Study
Arm/Group | Asthmatic Subjects | Without Asthma
Started | 12 | 14
Completed | 12 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Asthmatic Subjects | Without Asthma | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Continuous [Mean (Full Range); unit: years] | 24.1 [19 to 39] | 21.9 [20 to 27] | 22.9 [19 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 14 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 10 | 14 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Total IgE level [Geometric Mean (Full Range); unit: International Units/ml] | 1239 [596 to 4692] | 14 [2.4 to 42.5] | 110 [2.4 to 4692]
Negative serum antibody to Rhinovirus-16 [Count of Participants; unit: Participants] | 12 | 14 | 26

OUTCOME MEASURES:

1. Primary Outcome: Airway Symptom Scores Experienced by Subjects During the 1st 4 Days of the Infection
Description: The primary endpoint will be based on the comparison of cumulative lower respiratory tract symptom scores (CLRTS) in the asthmatic subjects compared to the non-asthmatic subjects over the first 4 days of acute infection. The symptoms evaluated daily included wheeze, chest tightness, shortness of breath, and cough. Symptom scores, including wheeze, shortness of breath, and chest discomfort were recorded by subjects twice daily. Each symptom was scored on a scale of 1-3. Therefore, the total maximum (worst) score for a day would be 24. The scores recorded daily could range from 0 to 24.
Time Frame: 4 days
Population: One asthmatic subject completed the study, but was dropped according to protocol because that subject acquired a cold after enrollment, but before rhinovirus inoculation. One subject without asthma was dropped according to protocol, because they did not develop a cold after inoculation with rhinovirus.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Asthmatic Subjects | Without Asthma
Number analyzed (Participants) | 11 | 13
units on a scale | 8.72 [1.55 to 15.91] | 2.77 [0.22 to 5.32]
Statistical Analysis 1: Comparison: Asthmatic Subjects vs Without Asthma; Test type: Superiority; p = 0.049, Negative binomial regression

2. Secondary Outcome: Airway Symptom Scores Experienced by Subjects During the 1st 4 Days of the Infection Evaluated Without Cough.
Description: Symptom scores, including wheeze, shortness of breath, and chest discomfort were recorded by subjects twice daily. Each symptom was scored on a scale of 1-3. Therefore, the total maximum (worst) score for a day would be 18. The scores recorded daily could range from 0 to 18.
Time Frame: 4 days
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Asthmatic Subjects | Without Asthma
Number analyzed (Participants) | 11 | 13
units on a scale | 6.09 [0.47 to 11.71] | 0.08 [0 to 0.24]
Statistical Analysis 1: Comparison: Asthmatic Subjects vs Without Asthma; Test type: Superiority; p < 0.001, Negative binomial regression

ADVERSE EVENTS:
Time Frame: 5 years
Description: Collection of adverse events is described in our protocol reviewed and approved by our IRB and the NIH.
Arm/Group | Asthmatic Subjects | Without Asthma
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/14
Other Adverse Events (participants affected / at risk) | 2/12 | 1/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asthmatic Subjects (N=12) | Without Asthma (N=14)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) — One subject developed a neutropenia count consistent with an adverse event (< 1500 cells/mm3).
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Symptoms consistent with Allergic Rhinitis developed in one asthmatic during the one week run-in period. The subject tested negative for virus during the run-in period.
Upset stomach (Gastrointestinal disorders) | 1 (1) | 0 (0) — One asthmatic developed an upset stomach (lasting a few hours) following the virus challenge. This was transient and resolved without intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-18): https://cdn.clinicaltrials.gov/large-docs/72/NCT02111772/Prot_SAP_000.pdf